CLINICAL TRIAL: NCT03490552
Title: RNA Sequencing Analysis in Large Vessel Occlusion Stroke DATA Bank (RNASA-LVOSB), the Futuristic Finger Print Recognition of Stroke Source
Brief Title: RNA Sequencing Analysis in Large Vessel Occlusion Stroke DATA Bank
Acronym: RNASA-LVOSB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Society of Minimally Invasive Neurological Therapeutic Procedures (Network)
Collaborators: Pakistani Society of Neuroradiology (Other); Middle east North Africa Stroke & interventional Neurotherapies Organization (Unknown); Egyptian Stroke Society (Other); African Academy of neurology (Unknown); Egyptian Society for Progenitor Cell Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: MENA-SINO-T001; MENASINO-001 (Other: MENA-SINO)
Record Dates: First submitted 2018-03-26; First posted 2018-04-06 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-03

CONDITIONS: Stroke, Acute; Thrombosis
MeSH Terms: conditions — Stroke; Thrombosis | interventions — Sequence Analysis, RNA

STUDY DESIGN:
Intervention Model Description: A double blind, randomized, controlled investigational study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Sham Comparator): include clots which have been extracted by mechanical thrombectomy and with definite stroke etiology and submitted to the RNA analysis in blinded coded label .
  Interventions: Procedure: mechanical thrombectomy
- group B (Experimental): include all clots which have been extracted by mechanical thrombectomy and with unknown stroke etiology and submitted to RNA analysis in cryptogenic label.
  Interventions: Procedure: mechanical thrombectomy

INTERVENTIONS:
Procedure: mechanical thrombectomy — Mechanical thrombectomy whatever it type ( SRT , ASPT or Mixed )will be used to extract the thrombi from stroke causing occlusion to be preserved biologically for genomic lab. transfer to be processed by RNA sequencing analysis technique for identifying markers for its composition pointing to its source.
  Other Names: RNA Sequencing Analysis

SUMMARY:
Introduction: the source of embolic stroke , in thrombotic embolism , is of unknown origin in 30-40% of cases. Fortunately , Mechanical thrombectomy provide a direct method to retrieve the stroke-incriminated clots from stroke patients for possibility of exo-autopsy analysis.

DETAILED DESCRIPTION:
Introduction: the source of embolic stroke , in thrombotic embolism , is of unknown origin in 30-40% of cases. Fortunately , Mechanical thrombectomy provide a direct method to retrieve the stroke-incriminated clots from stroke patients for possibility of exo-autopsy analysis.

Aim of the study : collecting stroke-incriminated clots from definite known etiological sources, could build a matchable markers database (MMD) to identify the source of cryptogenic embolism in the near-future. Identification of that markers is done by novel RNA sequencing technology to identify the clot composition in direct way.

Methodology: This is a prospective REB-approved study of acute LVO ischemic stroke in patients receiving mechanical thrombectomy at a multiple centers . Immediately after thrombi will be retrieved by mechanical thrombectomy, they will be placed in RNA stabilization and storage solution (RNAlater). Each sample will be extracted for total RNA by the one approved regional university's Human Genomics lab using a standard protocol. NanoDrop Microvolume Spectrophotometers and Fluorometer will be used for RNA quantification.

Thrombi weight will be recorded among other patient data , risk factors , procedural data, usage of adjunctive drugs and macroscopic morphology of each clot . Pearson correlation was used for correlation analysis.

all clots will be handled in double blinded control manner ; where clots analysis will be divided into 2 groups where Group A : include clots with definite stroke etiology and submitted to the RNA analysis in blinded coded label .

Group B: include all clots with unknown stroke etiology and submitted to RNA analysis in cryptogenic label .

the trial will be conducted over 4 years period from 2018 to 2022, with expected sample size of 350 cases with 7 : 3 ratio of enrollment in both groups ( a, b).

all analysis will be re-audited in central genome analysis lab of Alexandria University .

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature
2. Age ≥ 18 to < 86 years
3. Clinical signs consistent with an acute ischemic stroke
4. Neurological deficit with a NIHSS of ≥ 8 and < 30
5. Patient is eligible for intravenous thrombolysis
6. Patient is eligible for endovascular treatment
7. Randomization no later than 4 hours 15 minutes after stroke symptom onset and initiation of IV t-PA must be started within 4 hours 30 minutes of stroke symptoms onset (onset time is measured from the time when the subject was last seen well)
8. Occlusion (TICI 0-1) of the intracranial internal carotid artery (ICA), the M1 segment of the middle cerebral artery (MCA), or both confirmed by CT or MR angiography, accessible for MT
9. Core-infarct volume of Alberta Stroke Program Early CT Score (ASPECTS) greater than or equal to 6 (≥6) based on baseline CT or MR imaging (MRI)

Exclusion Criteria:

1. Acute intracranial hemorrhage
2. Any contraindication for IV t-PA
3. Pre-treatment with IV t-PA
4. In-hospital stroke
5. Pregnancy or lactating women. A negative pregnancy test before randomization is required for all women with child-bearing potential.
6. Known (serious) sensitivity to radiographic contrast agents, nickel, titanium metals, or their alloys
7. Known current participation in a clinical trial (investigational drug or medical device)
8. Renal insufficiency as defined by a serum creatinine > 2.0 mg/dl (or 176.8 µmol/l) or glomerular filtration rate (GFR) < 30 mL/min or requirement for hemodialysis or peritoneal dialysis
9. Severe comorbid condition with life expectancy less than 90 days at baseline
10. Known advanced dementia or significant pre-stroke disability (mRS score of ≥2)
11. Foreseeable difficulties in follow-up due to geographic reasons (e.g. patients living abroad)
12. Comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.
13. Subject currently uses or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day).
14. Known history of arterial tortuosity, pre-existing stent, other arterial disease and/or known disease at the femoral access site that would prevent the device from reaching the target vessel and/or preclude safe recovery after MT
15. Radiological confirmed evidence of mass effect or intracranial tumor (except small meningioma)
16. Radiological confirmed evidence of cerebral vasculitis
17. CTA or MRA evidence of carotid artery dissection
18. Evidence of additional distal intracranial vessel occlusion in another territory (i.e. A2 segment of anterior cerebral artery or M3, M4 segment of MCA) on initial NCCT/MRI or CTA/MRA

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Mrs | 30 days
  Modified ranking scale

SECONDARY OUTCOMES:
Sensitivity & Specificity | 4 years
  match sensitivity more than 90 % and Specificity more than 80%

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University , School of medicine , Neurology Department, Neurovascular Unit, Alexandria, Egypt